CLINICAL TRIAL: NCT06815809
Title: Floor-hugging Intervention: Managing Fear of Falling Through Floor Exposure and Developing After-fall Contingency
Acronym: Floor-HI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karlstad University (Other)
Responsible Party: Principal Investigator, Shashank Ghai, Associate Senior Lecturer, Karlstad University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2024-07271-01
Record Dates: First submitted 2025-01-31; First posted 2025-02-07 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Fear of Falling; Balance Changes; Healthy
Keywords: Fear of falling; Balance assessment; After fall contingency

STUDY DESIGN:
Intervention Model Description: This study will use a sequential design with multiple pre- and post-assessments. Participants will be evaluated at four time points: baseline (week 0), pre-intervention (week 3), post-intervention (week 6), and follow-up (week 9).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Floor-HI intervention (Experimental): In the Floor-HI intervention arm the participants will undergo a 3-week training, where training is performed thrice a week during a 1-hour session. The training is conducted in three systematic steps mentioned as following:
  1. Positioning on the floor: Participants assume a position on the floor, using the backward chaining method.
  2. Floor hugging: Participants will assume a position on the floor, which may include supine, prone, side-lying, or semi-prone/supine poses. They will be encouraged to simulate a fall scenario by observing their surroundings while engaging in deep breathing exercises.
  3. Getting back up from the floor: Participants will learn strategies to recover from a fall, tailored to their individual balance capabilities i.e., getting back up using supported furniture or without any support.
  The interventions are performed on printed surfaces that are attached to sports mat. These printed surfaces mimic high fall risk surfaces such as wet, icy, or snowy surfaces.
  Interventions: Behavioral: Floor-HI (intervention combines floor exposure with floor rise strategies)

INTERVENTIONS:
Behavioral: Floor-HI (intervention combines floor exposure with floor rise strategies) — Floor HI training consists of the following three systematic steps
  1. Positioning on the floor: Participants are first taught the backward chaining method. This technique involves using nearby furniture as support to move from an upright position to a kneeling position, through prone and side lying positions, and finally to a supine position.
  2. Ground hugging: In this phase, participants will assume a position on the floor. They are encouraged to simulate a fall scenario by observing their surroundings while using relaxation techniques. This includes deep breathing exercises.
  3. Getting up from the floor: The final phase focuses on teaching participants techniques to recover from a fall, tailored to their individual balance abilities.
  The intervention is carried out on printed surfaces that mimic high fall risk surfaces such as icy, cluttered, wet surfaces.

SUMMARY:
Fear of falling is a major public health problem and is characterized by a lack of confidence in one's ability to maintain balance and prevent falls. The fear can range from reasonable precautions to avoid slippery surfaces to an overwhelming fear that prevents people from performing everyday activities. Several factors contribute to this fear, including physical, psychological, social and environmental factors. These factors can not only lead to an increased tendency to fall, but also to increased anxiety, depression and social isolation, which can ultimately impair the individual's physical and mental health. Current approaches to help have only limited or moderate success, often because they do not take into account how the environment affects people's relationship with the floor.

For example, in urbanized societies, people spend less time in contact with the floor, which may have led to an individual's perception of the floor changing. This connection is not only physical, but can also involve a lack of mental and sensory familiarity. Without regular interaction with the floor in different positions, the individual may feel insecure or unfamiliar with the floor. This unfamiliarity can increase anxiety and encourage hypervigilant behavior that can lead to a fear of falling. Similarly, unfamiliarity with the floor can also contribute to a person's ability to respond effectively to a fall, often leaving the person unsure of what steps to take next.

The Floor-Hugging Intervention (Floor-HI) is a new intervention that can address these issues. The intervention consists of three main parts: learning how to get down on the floor, familiarizing oneself with the floor, and learning how to get back up. In the first part, participants learn how to lie down on the floor using evidence-based methods. The participant then practices lying on the floor to become more comfortable and less anxious. By repeatedly practicing lying on the floor in a safe environment, the intervention aims to break the connection between the floor and the fear associated with it, while promoting a more positive and confident mindset.

The third part of Floor-HI is to teach strategies for getting up from the floor. This is important to help participants gain the confidence and physical strength to recover from falls. Participants are given practice in different ways to get up, first with the help of furniture and then without assistance. The training aims not only to improve participants' physical abilities but also their confidence in dealing with falls.

Each session of the Floor HI programme is designed to last 1 hour and to be performed three times a week for three weeks. The training would be divided equally between getting used to the floor and learning to stand up. The results of the programme would be evaluated by assessing its impact on participants' fear of falling, static and dynamic balance, fall frequency, ability to get up from the floor and general quality of life. In addition, the acceptability of the intervention and any adverse events occurring as a result of participation in the intervention will also be collected. In conclusion, Floor-HI can be a good way to manage the fear of falling by focusing on both mental and physical aspects, which can ultimately help people to live more active and fulfilling lives.

DETAILED DESCRIPTION:
Background Fear of falling (FoF) is a serious public health problem affecting healthy and patient populations worldwide. It can range from a healthy caution that leads individuals to avoid environmental hazards such as icy, slippery roads or wet surfaces, to a disabling fear that forces them to stay at home, limiting their mobility and participation in activities of daily living. Several factors contribute to the development of FoF, including physical, cognitive, psychological, social and environmental influences. For example, in older adults, age-related declines in strength, sensation and cognitive function increase the risk of falling, which ultimately increases the FoF. Similarly, environmental factors such as icy winter conditions, particularly in Scandinavia, have been shown to increase FoF, not only in older adults but also in middle-aged and younger populations. FoF leads to self-imposed avoidance behaviors, meaning that individuals suffering from FoF voluntarily restrict their own mobility, which further worsens their health outcomes, increases their social isolation and reduces their overall quality of life. Ironically, this avoidance behavior, which is intended to prevent falls, has been reported to increase the risk of falling.

Despite the availability of interventions to reduce FoF, their effectiveness remains limited. One possible explanation is the lack of focus on the design of the environment, particularly on how individuals interact with the floor itself. In urbanized societies, direct contact with the floor through activities such as sitting, lying down or kneeling is rare. This lack of engagement can create a sense of unfamiliarity, similar to the discomfort a European might feel when eating with chopsticks in Asia, or a Swedish driver navigating left-hand traffic in the UK. Both examples illustrate how unfamiliarity with a task can lead to psychological uncertainty. For individuals with limited exposure to floor-based activities, this disconnect may similarly exacerbate psychological uncertainty about the floor and managing falls, intensifying FoF. Likewise, reduced engagement with floor-based activities in urbanized societies might also lead to deconditioning of the muscular strength and coordination needed to recover from falls. This could explain why adults who are do not know how to get back up after a fall experience heightened FoF.

These explanations are consistent with the uncertainty and anticipation model, which suggests that uncertainty about potential threats - such as falling - can increase threat expectancy. This overestimation of the risks associated with falling may in turn lead to maladaptive behaviors, including hypervigilance, avoidance, biased attention and poor updating of associative learning, all of which may contribute to increased FoF (10). Addressing this multifaceted problem therefore requires interventions that address underlying causes, such as limited ground exposure and inadequate post-fall recovery strategies, to mitigate the development of FoF.

The Floor Hugging Intervention (Floor-HI) is one such program that has been developed along these lines and may prove to be a potentially beneficial approach to alleviating FoF. The program comprises two main components: one aimed at enhancing familiarity with the floor and the other focused on developing post-fall strategies. Here, the first component of the Floor-HI, which deals with floor exposure, is based on emotional processing theory and allows for confrontation with the uncertainty of the floor and falls by asking individuals to lie on the floor in various positions while imagining that they have fallen. The act of spending time on the floor and imagining a fall in a safe environment is intended to create cognitive dissonance that can reshape and update fear structures to reduce the FoF. The second component of Floor-HI, which involves teaching individuals' strategies for getting back up after a fall, is intended to further empower individuals by increasing their self-efficacy in coping with falls, thereby further reducing the uncertainty (i.e. lack of post-fall contingencies) that also contributes to the development of FoF.

An innovative feature of Floor-HI is the use of printed surfaces that simulate high-risk environments such as icy, snowy, wet and cluttered surfaces, allowing participants to train in environments that reflect real-world challenges. This environmentally relevant approach ensures that training remains ecologically salient, safe while preparing individuals for potential hazards in a controlled and engaging manner. The program also addresses a critical gap in current government guidelines, which focus primarily on ground level strategies that rely on furniture for support. Such strategies may not be applicable in outdoor or unsupported environments. Floor-HI takes a personalized approach, allowing participants to choose between supported and unsupported floor-rising techniques based on their physical abilities.

Floor-HI Steps

Floor HI training consists of three systematic steps. In the first phase, participants assume a position on the floor. The second phase simulates a fall scenario. Finally, the individual regains an upright position using a supported or unsupported floor-rise strategy. The detailed steps are described below:

1. Positioning on the floor: Participants will initially be taught the backward chaining method, an evidence-based strategy for safely transitioning to the floor. This technique will involve using nearby furniture for support to move from an upright stance to a kneeling position, progressing through prone and lateral recumbent positions before ultimately assuming a supine posture.
2. Floor hugging: In this phase, participants will adopt a position on the floor, which may include supine, prone, side-lying, or semi-prone/supine poses. They will be encouraged to simulate a fall scenario by observing their surroundings while engaging in relaxation techniques. This will include practicing deep breathing exercises and listening to calming music to reduce anxiety.
3. Getting back up from the floor: The final phase will focus on teaching participants techniques to recover from a fall, tailored to their individual balance capabilities.

   * For individuals with poor balance, the forward chaining method will be employed, essentially reversing the backward chaining process. This step-by-step approach will transition from a supine position to side-lying, then to half-sitting, prone kneeling, high kneeling, half-kneeling, and finally to stride standing, with support from assistive furniture.
   * For individuals with good balance, such as young or middle-aged participants an approach which does not rely on the use of assistive furniture will be used. The approach would consist of seven key components: lying, initiating, positioning, supporting, elevation, stabilization, and transitioning to a standing posture.

The Floor-HI program has been thoughtfully designed in alignment with the biopsychosocial model of the International Classification of Functioning, Disability, and Health. This model emphasizes the interplay between biological, psychological, and social factors in promoting overall well-being. It is hypothesized that Floor-HI training will reduce the uncertainty associated with floor exposure and post-fall scenarios, thereby alleviating psychological distress. Moreover, the program is expected to enhance balance confidence and self-efficacy in managing falls, which could contribute to improved social well-being for participants. Physical benefits, such as improved static and dynamic balance and mobility, are also anticipated as participants build strength and coordination through repeated practice of floor-rising strategies.

To comprehensively evaluate the impact of the Floor-HI intervention on mobility and well-being, a thorough assessment is required. This includes examining its effects on FoF, balance ability, floor-rising ability, fall frequency, and quality of life. Additionally, understanding the program's implementation is essential. Evaluating participant acceptability and identifying any potential adverse events associated with Floor-HI will provide valuable insights for future optimization of the intervention.

Research questions

Primary question:

1. To evaluate the influence of Floor-HI on FoF in adults.

   Secondary questions:
2. To evaluate the influence of Floor-HI on postural stability, turn capacity, floor rising ability, fall incidences, and health-related quality of life.
3. To evaluate the acceptability of the Floor-HI.
4. To evaluate potential adverse events related to the Floor-HI.

Study design This study will use a sequential design with multiple pre- and post-assessments. Participants will be evaluated at four time points: baseline (week 0), pre-intervention (week 3), post-intervention (week 6), and follow-up (week 9). The strength of this design lies in its ability to incorporate a built-in control period. The initial 3-week interval between baseline and pre-intervention, during which participants will not undergo training, serves as a control period to assess the effectiveness of the Floor-HI intervention. Additionally, the follow-up assessment between weeks 6 and 9 will help determine whether the benefits gained from the 3-week Floor-HI training are retained over time.

Participants: Healthy adults (18 to 64 years) will be recruited for the study. The inclusion criteria for participation will be: i) adults with intact cognitive function (Montreal Cognitive Assessment score ≥ 26 out of 30); ii) adults who are functionally independent and able to perform activities of daily living without assistance; iii) adults who are not receiving concomitant balance training; iv) adults who can speak and understand either Swedish or English.

Sample size: The sample size calculation is based on the study's primary outcome, the Falls Efficacy Scale-International. According to the literature, a Minimal Clinically Important Difference of at least 5.5 points on the falls efficacy scale-international is considered significant from the patient's perspective. To ensure 90% statistical power, with an alpha error of 0.05 and assuming a medium effect size (Cohen's d = 0.50), the study requires a sample size of 44 participants. Accounting for an anticipated dropout rate of approximately 10%, the recruitment target is set at 48 participants.

Assessment: The efficacy of Floor-HI will be evaluated using the following tools:

1. FoF: FoF will be assessed using the Falls Efficacy Scale-International, a 16-item scale that measures concerns about falling during various activities. Participants will rate their level of concern on a 4-point Likert scale. Scores range from 16 to 64, with higher scores indicating a greater FoF.
2. Floor rising ability: Floor-rising ability will be assessed using the Sit-to-Stand Test, which measures the ability to sit and rise from the floor with minimal support. The test is scored from 0 to 10, with points deducted for the use of support or unstable movements. Higher scores indicate a better ability to rise from the floor.
3. Postural stability: Postural stability will be assessed using the Mini Balance Evaluation System Test, a 14-question tool that measures balance in several areas. Each question is scored from 0 to 2, with higher total scores (up to 28) indicating better balance.
4. Turning ability: Turning ability will be assessed using the 360° Turn Test, which evaluates dynamic balance. Participants will be asked to complete a full circle turn, with the time and/or number of steps taken recorded.

   Evaluated at four time points: baseline (week 0), pre-intervention (week 3), post-intervention (week 6), and follow-up (week 9).
5. Health-related quality of life: The 36-item RAND Health Survey will be used to assess health-related quality of life across eight health domains.
6. Fall incidence: Participants will record daily falls in a diary, noting the cause, location, and outcome of each fall.
7. Acceptability of the intervention: Acceptability will be assessed using the Theoretical Framework of Acceptability questionnaire, which evaluates participants' perceptions of the intervention based on seven constructs, including efficacy and self-efficacy.
8. Adverse events: Adverse events will be documented using the National Institute on Aging Adverse Event Form, recording any adverse events experienced by participants during the study role.

Ethical approval An ethical approval has been received for the project (2024-07271-01).

ELIGIBILITY:
Inclusion Criteria:

* Participants must be healthy adults between the ages of 18 and 64.
* Participants must be fluent in either Swedish or English.
* Participants must have a Montreal Cognitive Assessment (MoCA) score of 23 or higher.
* Participants must be able to perform activities of daily living independently.

Exclusion Criteria:

* Participants with neurological diseases (e.g., stroke, Parkinson's disease, multiple sclerosis, traumatic brain injury, etc.).
* Participants with musculoskeletal disorders (e.g., rheumatoid arthritis, sprains, strains, etc.).
* Participants with severe cognitive impairments (Montreal Cognitive Assessment score < 23).
* Participants with psychiatric disorders (e.g., bipolar disorder, schizophrenia).
* Participants currently involved in any other exercise-based interventions that involves prolonged floor contact (e.g., yoga, martial arts, dance).

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-02-11 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Falls Efficacy Scale-International | Evaluated at four time points: baseline (week 0), pre-intervention (week 3), post-intervention (week 6), and follow-up (week 9).
  Fear of falling will be evaluated using the 16-item Falls Efficacy Scale-International. This scale measures fear of falling during daily activities, making it suitable for active adults. Additionally, it incorporates the social aspects of this fear and has demonstrated strong measurement properties, even across different cultural settings.

SECONDARY OUTCOMES:
Sitting rising test | Evaluated at four time points: baseline (week 0), pre-intervention (week 3), post-intervention (week 6), and follow-up (week 9).
  The Sitting-Rising Test is an untimed assessment that will be used to evaluate an individual's ability to rise from the floor. This 5-point test measures both independence (i.e., ability to rise without support) and stability (as reported by the clinician). It has been proven to be responsive, reliable, and valid. During the test, one point is deducted each time the participant uses support to lower themselves or stand up, and 0.5 points are subtracted if the clinician observes instability during the movement.
Mini-BESTest | Evaluated at four time points: baseline (week 0), pre-intervention (week 3), post-intervention (week 6), and follow-up (week 9).
  The Mini-BESTest will be used to evaluate the impact of the Floor-HI program on both static and dynamic balance. This comprehensive assessment examines various aspects of balance control, including anticipatory postural adjustments, reactive responses, sensory integration, dynamic gait, stability limits, trunk stability, dual-task performance, and sitting balance. It is recognized for its high sensitivity, reliability, and validity in detecting balance impairments. The Mini-BESTest consists of 14 items, each scored from 0 to 2, with a maximum possible score of 28, where higher scores indicate better balance.
360° Turn Test | Evaluated at four time points: baseline (week 0), pre-intervention (week 3), post-intervention (week 6), and follow-up (week 9).
  The 360° Turn Test is a clinical tool used to assess dynamic balance and turning ability. In this test, an individual is instructed to perform a full 360° turn in either direction. The assessment is based on the time taken and/or the number of steps required to complete the turn. A faster completion time and fewer steps indicate better dynamic balance.
36-item RAND Health Survey | Evaluated at four time points: baseline (week 0), pre-intervention (week 3), post-intervention (week 6), and follow-up (week 9).
  The 36-Item RAND Health Survey is a self-reported questionnaire designed to assess an individual's health-related quality of life.The questionnaire evaluates eight key health domains: physical functioning, role limitations due to physical health problems, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems, and mental health. Each domain is scored on a scale from 0 to 100, with higher scores indicating better health status and quality of life.
Fall incidence (Fall diary) | Self-recorded by participants everyday from week 0 (baseline) to week 9 (follow-up) i.e., 63 days
  Participants will maintain a fall diary to document fall-related incidents during the 9-week study period. This diary will capture details such as the occurrence of a fall, the date it occurred, and the severity of any injuries sustained. Participants are expected to complete the diary at home and bring it to each assessment session (weeks 3, 6, and 9) for the researcher to record any falls. At the final evaluation, participants will submit the completed diary to the researcher.
Theoretical Framework of Acceptability questionnaire | Evaluated at two time points: pre-intervention (week 3) and post-intervention (week 6).
  The acceptability of the intervention will be assessed using the Theoretical Framework of Acceptability questionnaire. The tool assesses participants' views of the intervention through seven key constructs: attitude, burden, ethics, intervention coherence, opportunity cost, perceived effectiveness and self-efficacy. Each construct is assessed using a set of items rated on a 5-point Likert scale, with higher scores overall indicating greater acceptability of the intervention.

OTHER OUTCOMES:
National Institute on Aging Adverse Event Form | Evaluated during each training session i.e., nine training sessions during the course of three weeks
  Before and after each training session, participants will be asked about any side effects they may experience, including fatigue, pain, discomfort, and other negative or unwanted effects. These responses will be recorded on the National Institute on Aging Adverse Event Form V2.0 to track any potential adverse events throughout the course of the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- RiskLab, Karlstad University, Karlstad, Värmland County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
The IPD sharing is undecided due to ethical considerations and data privacy concerns. In the ethics application it had been made clear that group aggregates would be shared to prevent recognition of participants identity through their data.

REFERENCES:
- [Background] Sekhon M, Cartwright M, Francis JJ. Development of a theory-informed questionnaire to assess the acceptability of healthcare interventions. BMC Health Serv Res. 2022 Mar 1;22(1):279. doi: 10.1186/s12913-022-07577-3. PMID 35232455
- [Background] Ohlsson-Nevo E, Hiyoshi A, Noren P, Moller M, Karlsson J. The Swedish RAND-36: psychometric characteristics and reference data from the Mid-Swed Health Survey. J Patient Rep Outcomes. 2021 Aug 4;5(1):66. doi: 10.1186/s41687-021-00331-z. PMID 34347192
- [Background] Dite W, Temple VA. Development of a clinical measure of turning for older adults. Am J Phys Med Rehabil. 2002 Nov;81(11):857-66; quiz 867-8. doi: 10.1097/00002060-200211000-00010. PMID 12394998
- [Background] Potter K, Brandfass K. The Mini-Balance Evaluation Systems Test (Mini-BESTest). J Physiother. 2015 Oct;61(4):225. doi: 10.1016/j.jphys.2015.04.002. Epub 2015 Jun 1. No abstract available. PMID 26044345
- [Background] Araujo CGS, Castro CLB, Franca JFC, Araujo DS. Sitting-rising test: Sex- and age-reference scores derived from 6141 adults. Eur J Prev Cardiol. 2020 May;27(8):888-890. doi: 10.1177/2047487319847004. Epub 2019 May 1. No abstract available. PMID 31039614
- [Background] Halvarsson A, Stahle A. Psychometric properties of the Swedish version of the Falls Efficacy Scale-International for older adults with osteoporosis, self-reported balance deficits and fear of falling. Disabil Rehabil. 2018 Nov;40(22):2658-2661. doi: 10.1080/09638288.2017.1347210. Epub 2017 Jul 7. PMID 28687055
- [Background] Leonhardt R, Becker C, Gross M, Mikolaizak AS. Impact of the backward chaining method on physical and psychological outcome measures in older adults at risk of falling: a systematic review. Aging Clin Exp Res. 2020 Jun;32(6):985-997. doi: 10.1007/s40520-019-01459-1. Epub 2020 Jan 14. PMID 31939202
- [Background] Grupe DW, Nitschke JB. Uncertainty and anticipation in anxiety: an integrated neurobiological and psychological perspective. Nat Rev Neurosci. 2013 Jul;14(7):488-501. doi: 10.1038/nrn3524. PMID 23783199
- [Background] Feng C, Adebero T, DePaul VG, Vafaei A, Norman KE, Auais M. A Systematic Review and Meta-Analysis of Exercise Interventions and Use of Exercise Principles to Reduce Fear of Falling in Community-Dwelling Older Adults. Phys Ther. 2022 Jan 1;102(1):pzab236. doi: 10.1093/ptj/pzab236. PMID 34636923
- [Background] Lee D, Tak SH. A concept analysis of fear of falling in older adults: insights from qualitative research studies. BMC Geriatr. 2023 Oct 11;23(1):651. doi: 10.1186/s12877-023-04364-5. PMID 37821830
- [Background] Bjornstig U, Bjornstig J, Dahlgren A. Slipping on ice and snow--elderly women and young men are typical victims. Accid Anal Prev. 1997 Mar;29(2):211-5. doi: 10.1016/s0001-4575(96)00074-7. PMID 9088360
- [Background] Tinetti ME, Mendes de Leon CF, Doucette JT, Baker DI. Fear of falling and fall-related efficacy in relationship to functioning among community-living elders. J Gerontol. 1994 May;49(3):M140-7. doi: 10.1093/geronj/49.3.m140. PMID 8169336
- [Background] Xiong W, Wang D, Ren W, Liu X, Wen R, Luo Y. The global prevalence of and risk factors for fear of falling among older adults: a systematic review and meta-analysis. BMC Geriatr. 2024 Apr 5;24(1):321. doi: 10.1186/s12877-024-04882-w. PMID 38580924
- [Background] Ghai S, Ghai I. Floor-hugging Intervention: A Perspective on Floor Exposure and After-Fall Contingency Intervention. Adv Rehabil Sci Pract. 2024 Aug 22;13:27536351241271548. doi: 10.1177/27536351241271548. eCollection 2024 Jan-Dec. PMID 39184216